CLINICAL TRIAL: NCT06039072
Title: Clinical Observation on the Prognosis of Long-term Cardiac Function by Drug Withdrawal in Patients With Peripartum Cardiomyopathy With Cardiac Function Recovery
Brief Title: Clinical Observation of Long-term Cardiac Function Prognosis in Patients With PPCM Who Have Recovered Cardiac Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-2020(KS)-685
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples were collected for NT-proBNP values, routine blood tests (white blood cell count, hemoglobin, red blood cell count, platelet count, hematocrit), blood biochemistry (alanine aminotransferase, glutamine aminotransferase, urea nitrogen, creatinine, albumin, lipids, electrolytes, etc.), inflammatory markers (C-reactive protein, calcitonin), thyroid function (FT3, FT4, TSH, etc.), and markers of myocardial injury (troponin I, troponin T, creatine kinase isozymes, D-dimer, etc.), as well as genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects in the withdrawal group: Subjects received a combination of ACEI/ARB analogues, beta-blockers, MRA analogues, and diuretics during the standardized treatment phase, and after their cardiac function was restored, in order to avoid adverse effects on patients' cardiac function due to sudden withdrawal of drugs, the drugs were withdrawn according to a program to gradually stop the drug
  Interventions: Drug: Patients with cardiac function recovered for more than one year and discontinued were in the discontinuation group.
- Subjects in the continuing medication group: Subjects received a combination of ACEI/ARB analogues, beta-blockers, MRA analogues, and diuretics during the standardized treatment phase, and were continued on the original regimen after their cardiac function recovered

INTERVENTIONS:
Drug: Patients with cardiac function recovered for more than one year and discontinued were in the discontinuation group. — Among the patients with perinatal cardiomyopathy who were included in the study, their heart function returned to normal in 1 year after receiving standardized treatment, and then after another 1 year of standardized treatment to respect the patients' individual wishes, fully inform the patients of the relevant information and potential risks, including the possibility of deterioration of heart function after discontinuation of the medication, and only after obtaining the patients' informed consent and signing the informed consent form could they be included in the discontinuation group, and the rest were in the non-discontinuation group.
  Groups: Subjects in the withdrawal group

SUMMARY:
Peripartum cardiomyopathy (PPCM) is an idiopathic cardiomyopathy that occurs in late pregnancy and early postnatal period, which is mainly characterized by varying degrees of impaired ventricular systolic function and symptoms related to heart failure, and is a serious threat to maternal health. About 50% of patients can achieve complete recovery of cardiac function within 6 months after diagnosis with early standardized treatment, about 30%-40% of patients can have delayed recovery, and about 12.6% of patients have long-term impairment of cardiac function and poor prognosis. However, there are still controversies about whether and when to stop the drug after standardized treatment. The Chinese Society of Cardiovascular Disease of the Chinese Medical Association proposed in the Guidelines for the Diagnosis and Treatment of Dilated Cardiomyopathy in China that patients with PPCM should be considered for gradual withdrawal of the drug after at least 1 year of stabilization of cardiac structure and function recovery. And in the China Heart Failure and Diagnostic and Treatment Guidelines released in the same year, it is proposed that standardized heart failure therapy for patients with peripheral cardiomyopathy should be continued until at least 6 months after the left ventricular function has been fully recovered before gradual discontinuation of the drug. The American Heart Association's 2019 guidelines for perinatal cardiomyopathy remain skeptical about the timing of discontinuation, with some experts suggesting that the drug can be gradually discontinued 1-2 years after cardiac function has recovered, while others still recommend long-term use of the drug to avoid deterioration of cardiac function after discontinuation. At present, there is a lack of large-scale clinical studies on the effect of stopping standardized treatment on the long-term prognosis of PPCM patients, and clarifying whether PPCM patients can discontinue the drug and the timing of discontinuation is of great significance to the long-term prognosis of the patients and even to the rational allocation of the national healthcare resources as a whole.

DETAILED DESCRIPTION:
To clarify the effects of continuing standardized therapy and discontinuing standardized drug therapy on long-term cardiac function in patients with perinatal cardiomyopathy 1 year after cardiac function has been restored and stabilized, and to provide more theoretical and clinical bases for the therapeutic regimen of patients with perinatal cardiomyopathy after cardiac function is restored.

After diagnosis, patients received standardized heart failure treatment: according to the perinatal cardiomyopathy diagnosis and treatment guidelines of the Cardiovascular Disease Branch of the Chinese Medical Association and the American Heart Association, standardized heart failure treatment and symptomatic treatment were carried out according to the individualized differences of the patients, and for those who developed the disease in pregnancy, non-contraindicated medication was applied before delivery, and the appropriate mode of delivery was selected according to the gestation week and the cardiac function of the patient and the condition of the fetus, and the patients were given a comprehensive decision on the treatment plan by our hospital and the cardiologists and obstetricians of the collaborating hospitals. Cardiologists and obstetricians from our hospital and collaborating hospitals made comprehensive decisions on the treatment plan for the patients. The cardiologists and obstetricians of our hospital and the collaborating hospitals will make a comprehensive decision on the treatment plan of the patients. We will also assess whether the patients are suitable for breastfeeding, and choose non-contraindicated drugs and drugs with low milk concentration for breastfeeding, and standardize heart failure treatment as soon as possible after breastfeeding is finished; and for the non-breastfeeding patients, we will carry out the anti-heart failure treatment, applying the drugs such as ACEI/ARB, MRA and β-blocker as early as possible, and adjusting the dosage gradually according to the principle of individualization.

Treatment regimen for subjects in the discontinuation group: subjects received a combination of ACEI/ARBs, β-blockers, MRAs and diuretics during the standardized treatment phase, and after recovery of cardiac function, in order to avoid adverse effects on cardiac function caused by sudden withdrawal of medication, the medication was gradually discontinued in accordance with the protocol.

The completed case observation forms from each test center were retrieved after review by the supervisors and handed over to the main responsible unit (i.e., Qilu Hospital of Shandong University) for data processing. Data on the case report forms were entered in double copies by two persons, and the database was locked after verification to confirm that there were no errors. Measurement data were described by mean and standard deviation, and count data were described by number of cases and percentage. SPSS.23.0 statistical software was applied to statistically analyze the intention-to-treat set and the protocol-compliant set, respectively. The demographic characteristics of the enrolled cases in the two sets were first analyzed at baseline to examine the balance and comparability of the two sets. Then the effectiveness indicators and safety indicators of the two groups were compared.

For each index in the UCG, ECG, and a number of indicators such as blood pressure and heart rate between the experimental group and the control group; quantitative information was compared using the t-test for two-sample comparisons in a paired group design. At the same time, subgroup analyses were set up based on the NT-proBNP values of the patients and the time required for recovery of cardiac function, and univariate and multivariate statistical analyses were performed, and the primary endpoints were analyzed using the Kaplan-Meier survival curves with the log-rank-sum test, and the rank-sum tests for the group-designed two-sample comparisons were used for the NYHA classification and KCCQ scores. All statistical tests were two-sided, and a p-value less than or equal to 0.05 was considered statistically significant for the differences tested.

ELIGIBILITY:
Inclusion Criteria:

Perinatal cardiomyopathy patients aged 20-45 years who meet the diagnostic criteria for perinatal cardiomyopathy, i.e.: heart failure and left ventricular systolic hypoplasia occurring in the last trimester of gestation or 5 months postpartum; no previous history of heart failure and other etiologies that could explain the heart failure; impaired left ventricular function as indicated by cardiac ultrasound: LVEF <45% and/or FS <30% or left ventricular end-diastolic internal diameter ( LVEDd) > 5.0 cm; (ii) Those who have been diagnosed with perinatal cardiomyopathy and are now receiving standardized drug therapy, and whose cardiac function has not yet recovered, and whose enrollment time is not more than 1 year from the time of diagnosis.

Exclusion Criteria:

(i) Those with a previous history of severe organic valvular disease; (ii) Those with a previous history of diabetes mellitus, chronic hypertension and thyroid disease;

* Those with history of congenital heart disease, ischemic cardiomyopathy and other cardiomyopathies; ④ Those with severe infections and impaired liver and kidney functions (eGFR <30ml/min/1.73m2, or transaminases more than 5 times higher than the upper limit of normal values); ⑤ Those with previous persistent atrial, supraventricular or ventricular arrhythmia and have to be treated with anti-arrhythmic drugs for a long time; (vi) Those with serious adverse reactions and contraindications to heart failure therapeutic drugs.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Peripartum cardiomyopathy (PPCM) is an idiopathic cardiomyopathy that occurs in late pregnancy and the early postnatal period
Study Population: Source Clinical case collection of peripartum cardiomyopathy in multiple hospitals and recruitment of patients with peripartum cardiomyopathy，with recovery of cardiac function after standardized treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
deterioration in cardiac function within 1 year of the subgroup study | 1 year
  (i) a decrease in LVEF <10% and LVEF <50%; (ii) an increase in LVEDV of more than 10% and above the normal range; (iii) a 2-fold increase in NT-proBNP concentration of more than 400 ng/L; and (iv) the development of signs and symptoms of heart failure)

SECONDARY OUTCOMES:
patient cardiovascular accidents, rehospitalization-related adverse events | 1 year
  sustained arrhythmias, difficult-to-control hypertension, rehospitalization, and death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping ji, Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauersachs J, Konig T, van der Meer P, Petrie MC, Hilfiker-Kleiner D, Mbakwem A, Hamdan R, Jackson AM, Forsyth P, de Boer RA, Mueller C, Lyon AR, Lund LH, Piepoli MF, Heymans S, Chioncel O, Anker SD, Ponikowski P, Seferovic PM, Johnson MR, Mebazaa A, Sliwa K. Pathophysiology, diagnosis and management of peripartum cardiomyopathy: a position statement from the Heart Failure Association of the European Society of Cardiology Study Group on peripartum cardiomyopathy. Eur J Heart Fail. 2019 Jul;21(7):827-843. doi: 10.1002/ejhf.1493. Epub 2019 Jun 27. PMID 31243866
- [Background] Barasa A, Goloskokova V, Ladfors L, Patel H, Schaufelberger M. Symptomatic recovery and pharmacological management in a clinical cohort with peripartum cardiomyopathy. J Matern Fetal Neonatal Med. 2018 May;31(10):1342-1349. doi: 10.1080/14767058.2017.1317341. Epub 2017 May 2. PMID 28462600
- [Background] Biteker M, Ozlek B, Ozlek E, Cil C, Celik O, Dogan V, Basaran O. Predictors of early and delayed recovery in peripartum cardiomyopathy: a prospective study of 52 Patients. J Matern Fetal Neonatal Med. 2020 Feb;33(3):390-397. doi: 10.1080/14767058.2018.1494146. Epub 2018 Sep 27. PMID 29945487
- [Background] Davis MB, Arany Z, McNamara DM, Goland S, Elkayam U. Peripartum Cardiomyopathy: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jan 21;75(2):207-221. doi: 10.1016/j.jacc.2019.11.014. PMID 31948651
- [Background] Hilfiker-Kleiner D, Kaminski K, Podewski E, Bonda T, Schaefer A, Sliwa K, Forster O, Quint A, Landmesser U, Doerries C, Luchtefeld M, Poli V, Schneider MD, Balligand JL, Desjardins F, Ansari A, Struman I, Nguyen NQ, Zschemisch NH, Klein G, Heusch G, Schulz R, Hilfiker A, Drexler H. A cathepsin D-cleaved 16 kDa form of prolactin mediates postpartum cardiomyopathy. Cell. 2007 Feb 9;128(3):589-600. doi: 10.1016/j.cell.2006.12.036. PMID 17289576
- [Background] Pearson GD, Veille JC, Rahimtoola S, Hsia J, Oakley CM, Hosenpud JD, Ansari A, Baughman KL. Peripartum cardiomyopathy: National Heart, Lung, and Blood Institute and Office of Rare Diseases (National Institutes of Health) workshop recommendations and review. JAMA. 2000 Mar 1;283(9):1183-8. doi: 10.1001/jama.283.9.1183. PMID 10703781
- [Background] Halliday BP, Wassall R, Lota AS, Khalique Z, Gregson J, Newsome S, Jackson R, Rahneva T, Wage R, Smith G, Venneri L, Tayal U, Auger D, Midwinter W, Whiffin N, Rajani R, Dungu JN, Pantazis A, Cook SA, Ware JS, Baksi AJ, Pennell DJ, Rosen SD, Cowie MR, Cleland JGF, Prasad SK. Withdrawal of pharmacological treatment for heart failure in patients with recovered dilated cardiomyopathy (TRED-HF): an open-label, pilot, randomised trial. Lancet. 2019 Jan 5;393(10166):61-73. doi: 10.1016/S0140-6736(18)32484-X. Epub 2018 Nov 11. PMID 30429050
- [Background] Isogai T, Kamiya CA. Worldwide Incidence of Peripartum Cardiomyopathy and Overall Maternal Mortality. Int Heart J. 2019 May 30;60(3):503-511. doi: 10.1536/ihj.18-729. Epub 2019 Apr 25. PMID 31019181
- [Background] Otani K, Tokudome T, Kamiya CA, Mao Y, Nishimura H, Hasegawa T, Arai Y, Kaneko M, Shioi G, Ishida J, Fukamizu A, Osaki T, Nagai-Okatani C, Minamino N, Ensho T, Hino J, Murata S, Takegami M, Nishimura K, Kishimoto I, Miyazato M, Harada-Shiba M, Yoshimatsu J, Nakao K, Ikeda T, Kangawa K. Deficiency of Cardiac Natriuretic Peptide Signaling Promotes Peripartum Cardiomyopathy-Like Remodeling in the Mouse Heart. Circulation. 2020 Feb 18;141(7):571-588. doi: 10.1161/CIRCULATIONAHA.119.039761. Epub 2019 Oct 31. PMID 31665900
- [Background] Li W, Li H, Long Y. Clinical Characteristics and Long-term Predictors of Persistent Left Ventricular Systolic Dysfunction in Peripartum Cardiomyopathy. Can J Cardiol. 2016 Mar;32(3):362-8. doi: 10.1016/j.cjca.2015.07.733. Epub 2015 Aug 15. PMID 26586094
- [Background] Shani H, Kuperstein R, Berlin A, Arad M, Goldenberg I, Simchen MJ. Peripartum cardiomyopathy - risk factors, characteristics and long-term follow-up. J Perinat Med. 2015 Jan;43(1):95-101. doi: 10.1515/jpm-2014-0086. PMID 24887948